CLINICAL TRIAL: NCT07395726
Title: Impact of Platelet-Rich Fibrin on Periodontal Tissue Regeneration: A Randomized Controlled Trial
Brief Title: Impact of Platelet-Rich Fibrin on Periodontal Tissue Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Ahmed Abdullah, Dr, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21MDC1
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Periodontitis; Periodontal Intrabony Defects
Keywords: Platelet-Rich Fibrin; Periodontitis; Periodontal Regeneration; Probing Pocket Depth; Clinical Attachment Level
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Flap Debridement (Placebo Comparator): Participants assigned to this arm will undergo conventional open flap debridement (OFD) for the treatment of periodontal intrabony defects. The procedure involves flap elevation, thorough debridement of granulation tissue, root surface instrumentation, defect decontamination, and flap repositioning with suturing. Standard postoperative care and oral hygiene instructions will be provided.
  Interventions: Procedure: Open Flap Debridement
- Platelet-Rich Fibrin with Open Flap Debridement (Experimental): Participants assigned to this arm will receive autologous Platelet-Rich Fibrin (PRF) as an adjunct to conventional open flap debridement. PRF will be prepared from the participant's venous blood using centrifugation and placed directly into the periodontal defect prior to flap closure to promote tissue regeneration and enhance healing. All other surgical and postoperative procedures will be identical to the control group.
  Interventions: Procedure: Platelet-Rich Fibrin with Open Flap Debridement

INTERVENTIONS:
Procedure: Open Flap Debridement — Participants assigned to this arm will undergo conventional open flap debridement (OFD) for the treatment of periodontal intrabony defects. The procedure involves flap elevation, thorough debridement of granulation tissue, root surface instrumentation, defect decontamination, and flap repositioning with suturing. Standard postoperative care and oral hygiene instructions will be provided.
  Arms: Open Flap Debridement
Procedure: Platelet-Rich Fibrin with Open Flap Debridement — Participants assigned to this arm will receive autologous Platelet-Rich Fibrin (PRF) as an adjunct to conventional open flap debridement. PRF will be prepared from the participant's venous blood using centrifugation and placed directly into the periodontal defect prior to flap closure to promote tissue regeneration and enhance healing. All other surgical and postoperative procedures will be identical to the control group.
  Arms: Platelet-Rich Fibrin with Open Flap Debridement

SUMMARY:
The purpose of this research is to assess the efficacy of Platelet-Rich Fibrin (PRF) in the regeneration of periodontal tissues in patients suffering from periodontal disease. Periodontal disease is a chronic inflammatory disease that affects the gums and the bone supporting the teeth, which can eventually result in the loss of teeth if left untreated. Conventional periodontal treatment can control the infection and halt the progression of the disease but cannot reverse the loss of the supporting structures.

Platelet-Rich Fibrin is a biologic material derived from a small amount of the patient's own blood. It has growth factors that can potentially enhance healing and facilitate the regeneration of bone and soft tissues. In this randomized controlled clinical trial, patients will be randomly assigned to either conventional periodontal surgical treatment or conventional treatment along with PRF.

Over a predetermined follow-up period, clinical measurements like gum pocket depth, attachment levels, and radiographic bone changes will be assessed to see if PRF offers any extra advantages in tissue healing and regeneration. The results of this study could improve long-term oral health outcomes and periodontal disease treatment approaches.

DETAILED DESCRIPTION:
Periodontal disease is marked by the inflammation-mediated loss of the supporting structures of the teeth, leading to the formation of periodontal pockets, loss of clinical attachment, and resorption of the alveolar bone. The regenerative aspect of periodontal therapy aims at the replacement of these lost structures to improve the stability of the teeth and their functional status in the oral environment. Platelet-Rich Fibrin (PRF), an autologous platelet concentrate derived from the centrifugation of the patient's blood, is a fibrin matrix rich in growth factors that could potentially improve wound healing, angiogenesis, and bone regeneration.

The aim of this randomized controlled clinical trial is to assess the additional role of PRF when used in combination with conventional periodontal surgical therapy compared to conventional therapy alone in patients diagnosed with periodontal defects that require surgical treatment. The participants will be randomly assigned into two groups. The control group will undergo conventional periodontal surgical therapy, while the intervention group will undergo the same surgical therapy plus PRF. The procedures will be carried out according to standardized clinical protocols to ensure uniformity among the participants.

The clinical outcomes will be measured by changes in pocket depth, clinical attachment level, and other periodontal parameters. Radiographic analysis will also be conducted to evaluate bone fill and regenerative outcomes at specific intervals. The safety of the procedure will be continuously monitored, and since the PRF is autologous, the risk of immunologic reaction is minimal.

This study will offer high-quality evidence on the effectiveness of PRF as a regenerative tool in periodontal therapy and may help in making better clinical decisions in the treatment of periodontal defects.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years. Diagnosed with chronic periodontitis according to standard clinical criteria. Presence of periodontal intrabony defects suitable for surgical intervention. Probing pocket depth (PPD) ≥ 5 mm at the target site. Clinical attachment level (CAL) loss ≥ 3 mm at the target site. Good oral hygiene, with full-mouth plaque score < 25%.

Exclusion Criteria:

* Patients with systemic diseases that affect healing (e.g., uncontrolled diabetes, immunodeficiency).

Pregnant or lactating women. Current smokers or tobacco users. History of periodontal surgery at the target site within the last 12 months. Use of medications that interfere with wound healing (e.g., corticosteroids, bisphosphonates).

Allergies or contraindications to local anesthetics or components used in the study.

Active oral infections or untreated caries at or near the target site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-10-25 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Probing Pocket Depth (PPD) | Baseline to 6 months postoperatively.
  Probing pocket depth will be measured in millimeters using a calibrated periodontal probe at the selected defect sites. The outcome will be defined as the mean reduction in PPD from baseline to 6 months following surgery.

SECONDARY OUTCOMES:
Change in Clinical Attachment Level (CAL) | Baseline to 6 months postoperatively.
  Clinical attachment level will be assessed in millimeters using a standardized periodontal probe. The outcome will be defined as the mean gain in CAL from baseline to 6 months after treatment.
Percentage of Radiographic Bone Fill | Baseline to 6 months postoperatively.
  Bone regeneration will be evaluated using cone-beam computed tomography (CBCT). The percentage of bone fill within the periodontal defect will be calculated by comparing baseline and 6-month radiographic measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institute of Dentistry, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No
Many single-center clinical trials, especially in dentistry, do not share IPD publicly.
  Sharing IPD requires additional ethical approval, consent language, and data management plans.